CLINICAL TRIAL: NCT00320385
Title: A Randomized, Multicenter, Open-Label, Phase III Study of Lapatinib in Combination With Trastuzumab Versus Lapatinib Monotherapy in Subjects With HER2-positive Metastatic Breast Cancer Whose Disease Has Progressed on Trastuzumab-Containing Regimens
Brief Title: Lapatinib In Combination With Trastuzumab Versus Lapatinib Monotherapy In Subjects With HER2-positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EGF104900
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Results first posted 2011-11-30 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2015-04

CONDITIONS: Neoplasms, Breast
Keywords: lapatinib; GW572016; ErbB2; EGFR; ErbB1; MBC; FISH amplification; Metastatic Breast Cancer; dual tyrosine kinase inhibitor; Her-2/neu
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Lapatinib plus Trastuzumab (Experimental): Lapatinib 1000mg once daily in combination with trastuzumab 4mg/kg loading dose followed by 2mg/kg weekly
  Interventions: Drug: Lapatinib; Biological: Trastuzumab
- Arm 2: Lapatinib (Experimental): Lapatinib 1500mg once daily
  Interventions: Drug: Lapatinib

INTERVENTIONS:
Drug: Lapatinib — oral lapatinib once daily
  Other Names: Tyverb; Tykerb
Biological: Trastuzumab — IV trastuzumab 2mg/kg weekly after 4mg/kg loading dose
  Other Names: Herceptin
  Arms: Arm 1: Lapatinib plus Trastuzumab

SUMMARY:
This study will evaluate and compare the safety and efficacy of lapatinib in combination with trastuzumab versus lapatinib monotherapy in subjects with HER2-positive metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Female ≥18 years. Women of childbearing potential must have a negative serum pregnancy test at screening and must use an approved contraceptive method, if appropriate (for example, intrauterine device [IUD], birth control pills, or barrier device) beginning 2 weeks before the first dose of investigational product and for 28 days after the final dose of investigational product.
* Metastatic breast cancer, histologically/cytologically confirmed. If the disease is restricted to a solitary lesion, its neoplastic nature must be confirmed by cytology or histology.
* Subjects must have stage IV breast cancer whereby their disease has progressed in either the adjuvant or metastatic setting. Prior therapies must include, but are not limited to:
* Taxane-containing regimen for at least 4 cycles, or 2 cycles provided disease progression occurred while on taxane.
* Anthracycline-containing regimen for at least 4 cycles, or 2 cycles provided disease progression occurred while on anthracycline.
* Subjects must have documented progression following at least ONE trastuzumab plus cytotoxic chemotherapy or anti-hormonal regimen in the metastatic setting.
* Note: The most recent treatment must have contained trastuzumab, either alone or in combination with other therapy in the metastatic setting, and subjects must have progressed while on this regimen. Progression is defined as either new lesions or a ≥20% increase in the sum of longest diameter (LD) on the progression radiologic scan.
* Subjects must have archived tumor tissue available for testing.
* Documented amplification of the ErbB2 gene by fluorescence in situ hybridization (FISH) or documented overexpression of the ErbB2 protein by IHC in primary or metastatic tumor tissue. The IHC or FISH amplification may be documented by a local or central laboratory for randomization into the study. Subjects may be randomized on the basis of ErbB2 positivity by IHC 3+ overexpression or FISH amplification.
* Lesion eligibility is as follows:
* at least one measurable lesion(s) according to Response Evaluation Criteria in Solid Tumors [RECIST; Therasse, 2000], or
* bone-only disease.
* Note: Tumor lesions which are situated in a previously irradiated field, and have well-defined margins which are located in soft tissue will be defined as measurable disease.
* Subjects with stable CNS metastases defined as asymptomatic and off systemic steroids and anticonvulsants for at least 1 month. Treatment with prophylactic anticonvulsants is permitted, unless listed within the Prohibited Medications (Section 8.2).
* Radiotherapy if received within 2 weeks prior to initiation of investigational product to a limited area (e.g., palliative treatment for painful disease) other than the sole site of measurable disease is allowed; however, subject must have completed treatment and recovered from all treatment-related toxicities prior to administration of the first dose of investigational product.
* With the single exception of prior trastuzumab treatment, all prior chemotherapy, immunotherapy, biologic therapy, or surgery (except for minor surgical procedures) must be discontinued at least 3 weeks prior to the first dose of investigational product. Subjects must have recovered or stabilized sufficiently from treatment-related toxicities prior to administration of the first dose of investigational product.
* Bisphosphonate therapy for bone metastases is allowed; however, treatment must be initiated prior to the first dose of investigational product. Prophylactic use of bisphosphonates is permitted only for the treatment of osteoporosis.
* ECOG Performance Status of 0 to 2.
* Able to swallow and retain oral medication.
* Cardiac ejection fraction within institutional range of normal as measured by echocardiogram. MUGA scans will be accepted in cases where an echocardiogram cannot be performed or is inconclusive. Same modality used at baseline must be used for repeat assessments throughout study.
* Subject must have adequate organ function as defined in Table 1 :
* Table 1 (Definitions for Adequate Hematologic and Hepatic Function)
* SYSTEM (LABORATORY VALUES)
* Hematologic:
* ANC (absolute neutrophil count) (≥ 1x10^9/ L)
* Hemoglobin (≥ 9 g / dL)
* Platelets (≥75x10^9/ L)
* Hepatic
* Albumin (≥ 2.5 g / dL)
* Serum bilirubin (≤ 2 mg / dL)
* AST and ALT (≤ 3 x ULN without liver metastases) (≤ 5 xULN if documented liver metastases)
* Renal
* Serum Creatinine (≤1.5 mg / dL)
* OR -
* Calculated Creatinine Clearance1 (≥40 mL / min)
* Calculated by the Cockcroft and Gault Method.
* Subjects may continue anti-estrogen therapy only if treatment was initiated at least 1 month prior to the first dose of investigational product (IP). After randomization, no anti-hormonal therapy may be initiated.

Exclusion Criteria:

* Pregnant or lactating females.
* Prior therapy with an ErbB1 and/or ErbB2 inhibitor other than trastuzumab.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel. Subjects with ulcerative colitis are also excluded.
* History of other malignancy. However, subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
* Concurrent disease or condition that would make the subject inappropriate for study participation or any serious medical disorder that would interfere with the subject's safety.
* Unresolved or unstable, serious toxicity from prior administration of another investigational drug and/or of prior cancer treatment.
* Active or uncontrolled infection.
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
* Known history of uncontrolled or symptomatic angina, arrhythmias, or congestive heart failure.
* Known history or clinical evidence of leptomeningeal carcinomatosis.
* Concurrent cancer therapy (chemotherapy, radiation therapy, immunotherapy, biologic therapy).
* Concurrent treatment with an investigational agent or participation in another clinical trial.
* Used an investigational drug within 3 weeks or 5 half-lives, whichever is longer, preceding the first dose of investigational product.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to trastuzumab or lapatinib or their excipients.
* Have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2005-11; Primary Completion 2007-06 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (131):
- United States (82):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Sedona, Arizona
  - GSK Investigational Site, Highland, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Santa Rosa, California
  - GSK Investigational Site, Vallejo, California
  - GSK Investigational Site, Newark, Delaware
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Ocoee, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Niles, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Terre Haute, Indiana
  - GSK Investigational Site, Cedar Rapids, Iowa
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Robbinsdale, Minnesota
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Saint Joseph, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Montclair, New Jersey
  - GSK Investigational Site, Morristown, New Jersey
  - GSK Investigational Site, New Brunswick, New Jersey
  - GSK Investigational Site, Summit, New Jersey
  - GSK Investigational Site, Voorhees Township, New Jersey
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Cary, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Kettering, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Bryn Mawr, Pennsylvania
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Kingston, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, West Reading, Pennsylvania
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Beaumont, Texas
  - GSK Investigational Site, Bedford, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Denton, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Fredericksburg, Texas
  - GSK Investigational Site, Lewisville, Texas
  - GSK Investigational Site, Longview, Texas
  - GSK Investigational Site, McAllen, Texas
  - GSK Investigational Site, Mesquite, Texas
  - GSK Investigational Site, Midland, Texas
  - GSK Investigational Site, Odessa, Texas
  - GSK Investigational Site, Paris, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Salem, Virginia
  - GSK Investigational Site, Edmonds, Washington
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Vancouver, Washington
  - GSK Investigational Site, Yakima, Washington
  - GSK Investigational Site, Green Bay, Wisconsin
- Austria (2):
  - GSK Investigational Site, Salzburg
  - GSK Investigational Site, Vienna
- Bulgaria (2):
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Sofia
- Canada (2):
  - GSK Investigational Site, Laval, Quebec
  - GSK Investigational Site, Montreal, Quebec
- Croatia (2):
  - GSK Investigational Site, Split
  - GSK Investigational Site, Zagreb
- Czechia (2):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Prague
- GSK Investigational Site, Tampere, Finland
- Germany (17):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Coburg, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Fürstenwalde, Brandenburg
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Leer, Lower Saxony
  - GSK Investigational Site, Herne, North Rhine-Westphalia
  - GSK Investigational Site, Troisdorf, North Rhine-Westphalia
  - GSK Investigational Site, Velbert, North Rhine-Westphalia
  - GSK Investigational Site, Saarbrücken, Saarland
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
- Greece (2):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Neo Faliro
- Italy (6):
  - GSK Investigational Site, Bari, Apulia
  - GSK Investigational Site, Lecce, Apulia
  - GSK Investigational Site, Ravenna, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Rozzano (MI), Lombardy
  - GSK Investigational Site, Perugia, Umbria
- Poland (4):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- Spain (6):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Hospitalet de Llobregat (Barcelona)
  - GSK Investigational Site, Lleida
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santa Cruz de Tenerife
  - GSK Investigational Site, Valencia
- United Kingdom (3):
  - GSK Investigational Site, Huddersfield
  - GSK Investigational Site, Ipswich
  - GSK Investigational Site, London

REFERENCES:
- [Background] Wu Y, Amonkar MM, Sherrill BH, O'Shaughnessy J, Ellis C, Baselga J, Blackwell KL, Burstein HJ. Impact of lapatinib plus trastuzumab versus single-agent lapatinib on quality of life of patients with trastuzumab-refractory HER2+ metastatic breast cancer. Ann Oncol. 2011 Dec;22(12):2582-2590. doi: 10.1093/annonc/mdr014. Epub 2011 Mar 15. PMID 21406472
- [Background] Blackwell KL, Burstein HJ, Storniolo AM, Rugo HS, Sledge G, Aktan G, Ellis C, Florance A, Vukelja S, Bischoff J, Baselga J, O'Shaughnessy J. Overall survival benefit with lapatinib in combination with trastuzumab for patients with human epidermal growth factor receptor 2-positive metastatic breast cancer: final results from the EGF104900 Study. J Clin Oncol. 2012 Jul 20;30(21):2585-92. doi: 10.1200/JCO.2011.35.6725. Epub 2012 Jun 11. PMID 22689807

RESULTS

PARTICIPANT FLOW:
Groups:
- Trastuzumab + Lapatinib: Participants received Lapatinib 1000 milligram (mg) tablets orally daily 1 hour before or after breakfast along with Trastuzumab infusion at a loading dose of 4 milligrams/kilogram (mg/kg) body weight intravenously (IV) over 90 minutes on Day 1, followed by 2 mg/kg IV over 30 minutes weekly, in a 4 week cycle.
- Lapatinib: Participants received Lapatinib 1500 mg tablets orally daily 1 hour before or after breakfast.
Period: Overall Study
Arm/Group | Trastuzumab + Lapatinib | Lapatinib
Started | 148 | 148
Completed | 130 | 126
Not Completed | 18 | 22
Not completed — Lost to Follow-up | 7 | 10
Not completed — Withdrawal by Subject | 6 | 7
Not completed — Sponsor Terminated Study | 2 | 1
Not completed — Investigator Decision | 0 | 1
Not completed — Death | 1 | 2
Not completed — Serious Adverse Event | 1 | 0
Not completed — Withdrew Consent | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trastuzumab + Lapatinib | Lapatinib | Total
Number analyzed (Participants) | 148 | 148 | 296
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.1 (11.60) | 51.0 (10.40) | 51.5 (11.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 148 | 296
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 137 | 140 | 277
  African American/African Heritage | 6 | 5 | 11
  Asian | 2 | 3 | 5
  American Indian or Alaska Native | 1 | 0 | 1
  Native Hawaiian or other Pacific Islander | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from randomization until the first documented sign of disease progression or death due to any cause.
Time Frame: Baseline to disease progression or death due to any cause or 30 days after last dose (up to 216 weeks)
Population: Intent-to-Treat (ITT) Population: all randomized participants irrespective of whether or not they actually received study treatment. Only participants with progesterone receptor status were considered for evaluation.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Trastuzumab + Lapatinib | Lapatinib
Number analyzed (Participants) | 146 | 145
weeks | 12.0 [8.1 to 16.0] | 8.1 [7.6 to 9.0]
Statistical Analysis 1: Comparison: Trastuzumab + Lapatinib vs Lapatinib; Test type: Superiority or Other; p = 0.008, Log Rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.57 to 0.93] — The Pike estimator of the treatment hazard ratio based on the log-rank test was provided, together with a 95% confidence interval

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization until death due to any cause. For participants who did not die, OS was censored at the time of last contact.
Time Frame: Baseline to death or 30 days after last dose for the last participant (up to 216 weeks)
Population: ITT Population. Only participants with progesterone receptor status were considered for evaluation.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Trastuzumab + Lapatinib | Lapatinib
Number analyzed (Participants) | 146 | 145
weeks | 51.6 [42.9 to 57.3] | 39.0 [32.9 to 52.1]
Statistical Analysis 1: Comparison: Trastuzumab + Lapatinib vs Lapatinib; Test type: Superiority or Other; p = 0.106, Log Rank; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.53 to 1.07] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Overall Tumor Response (OR)
Description: OR was defined as the percentage of participants experiencing either a confirmed complete response (CR) or a confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.0. CR was defined as the disappearance of all lesions (target and/or non-target). PR was defined as at least a 30% decrease in the sum of the longest dimensions (LD) of target lesions taking as a reference the baseline sum LD, with non-target lesions not increased or absent.
Time Frame: Baseline to disease progression or death or discontinuation from study or 30 days after last dose (up to 216 weeks)
Population: ITT Population. Only participants with progesterone receptor status were considered for evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab + Lapatinib | Lapatinib
Number analyzed (Participants) | 146 | 145
percentage of participants | 10.3 | 6.9
Statistical Analysis 1: Comparison: Trastuzumab + Lapatinib vs Lapatinib; Test type: Superiority or Other; p = 0.460, Fisher Exact; Odds Ratio (OR) = 1.5, 95% CI 2-sided [0.6 to 3.9] — Responses were compared between treatment arms using stratified Fisher's exact tests

4. Secondary Outcome: Clinical Benefit Response (CBR)
Description: CBR: percentage of participants with confirmed CR or PR or stable disease (SD) for at least 24 weeks according to RECIST criteria. CR: disappearance of all lesions (target and/or non-target). PR: at least a 30% decrease in the sum of the LD of target lesions taking as reference baseline sum LD, with non-target lesions not increased or absent. SD: neither had sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD) in target lesions, taking as reference the smallest sum LD since treatment started; persistence of 1 or more non-target lesions.
Time Frame: Baseline to disease progression or death or discontinuation from study or 30 days after last dose (up to 216 weeks)
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab + Lapatinib | Lapatinib
Number analyzed (Participants) | 148 | 148
percentage of participants | 24.7 | 12.4
Statistical Analysis 1: Comparison: Trastuzumab + Lapatinib vs Lapatinib; Test type: Superiority or Other; p = 0.010, Fisher Exact; Odds Ratio (OR) = 2.2, 95% CI 2-sided [1.2 to 4.5] — Clinical Benefit was compared between treatment arms using stratified Fisher's exact tests

5. Secondary Outcome: Time to Response (TTR)
Description: TTR was defined as the time from randomization until the first documented evidence of CR or PR (whichever status was recorded first). TTR could not be analyzed because too few participants experienced a confirmed CR or PR.
Time Frame: Baseline until first documented evidence of CR or PR or 30 days after last dose (up to 216 weeks)
Population: ITT Population
Arm/Group | Trastuzumab + Lapatinib | Lapatinib
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Duration of Response (DR)
Description: DR was defined for the subset of participants who showed a confirmed CR or PR, as the time from the first documented evidence of CR or PR until the first documented sign of disease progression or death. Because of the low number of participants experiencing a confirmed response in both treatment arms, analysis for this outcome measure was not performed.
Time Frame: Time from first documented evidence of CR or PR until the first documented sign of disease progression or death or 30 days after last dose (up to 216 weeks)
Population: ITT Population
Arm/Group | Trastuzumab + Lapatinib | Lapatinib
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Time to Progression (TTP)
Description: TTP was defined as the interval between the date of randomization and the earlier of the date of disease progression or death due to breast cancer. Because this outcome measure was confounded by death due to other causes and was similar to PFS, it was not analyzed.
Time Frame: Baseline to disease progression or death or 30 days after last dose (up to 216 weeks)
Population: ITT Population
Arm/Group | Trastuzumab + Lapatinib | Lapatinib
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Breast (FACT-B) Scores at Week 4, Week 12, Week 16, Week 24, and Conclusion or Withdrawal From Study
Description: Quality of Life (QOL) was assessed using the FACT-B questionnaire, which was a 37-item (27 general and 10 breast cancer-specific questions) self-reporting instrument consisting of 5 dimensions: physical-, social/family-, emotional-, functional-well being, and a breast cancer subscale. Higher scores on the FACT-B scales indicate a higher QOL; each ranging from 0 (not at all) to 4 (very much). The score is transformed for FACT-B and results in a total score ranging from 0 to 144.
Time Frame: Baseline, Week 4, Week 12, Week 16, Week 24, and conclusion or withdrawal from study (up to Week 108)
Population: Safety Population: all randomized participants who received >=1 dose of investigational product. The Safety Population was based on the actual treatment received, if this differed from that to which the participant was randomized. Only participants whose overall item response rate was greater than 80% for the FACT-B total score were considered (n).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Trastuzumab + Lapatinib | Lapatinib
Number analyzed (Participants) | 137 | 137
scores on a scale
  Baseline, n=137, 137 | 98.7 (21.17) | 97.2 (21.85)
  Change at Week 4, n=101, 109 | -0.4 (11.52) | -0.6 (13.00)
  Change at Week 12, n=57, 51 | 1.5 (10.87) | -3.0 (12.54)
  Change at Week 16, n=42, 38 | -0.1 (13.34) | 0.4 (17.65)
  Change at Week 24, n=28, 28 | 1.3 (12.60) | -1.3 (15.67)
  Change at Conclusion/Withdrawal, n=63, 67 | -7.3 (15.48) | -8.0 (15.54)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from Baseline to conclusion or withdrawal from study; time from the first dose of treatment until 30 days after the last dose of study treatment (up to 216 weeks).
Description: SAEs and AEs were collected in the Safety Population, which consisted of all randomized participants who received at least one dose of investigational product, and was based on the actual treatment received, if this differed from that to which the participant was randomized.
Arm/Group | Trastuzumab + Lapatinib | Lapatinib
Serious Adverse Events (participants affected / at risk) | 40/149 | 24/146
Other Adverse Events (participants affected / at risk) | 140/149 | 132/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab + Lapatinib (N=149) | Lapatinib (N=146)
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Ejection fraction decreased (Investigations) | 7 | 1
Weight decreased (Investigations) | 0 | 1
Convulsion (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 0
Brain oedema (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 2
Cardiac failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Internal injury (Injury, poisoning and procedural complications) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab + Lapatinib (N=149) | Lapatinib (N=146)
Diarrhea (Gastrointestinal disorders) | 92 | 70
Nausea (Gastrointestinal disorders) | 42 | 41
Rash (Skin and subcutaneous tissue disorders) | 35 | 43
Fatigue (General disorders) | 33 | 29
Vomiting (Gastrointestinal disorders) | 22 | 26
Decreased appetite (Metabolism and nutrition disorders) | 20 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 14
Headache (Nervous system disorders) | 16 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 8
Asthenia (General disorders) | 11 | 10
Blood alkaline phosphatase increased (Investigations) | 11 | 5
Dyspepsia (Gastrointestinal disorders) | 10 | 11
Pyrexia (General disorders) | 10 | 7
Constipation (Gastrointestinal disorders) | 9 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 14
Aspartate aminotransferase increased (Investigations) | 9 | 3
Ejection fraction decreased (Investigations) | 9 | 1
Abdominal pain (Gastrointestinal disorders) | 8 | 7
Abdominal pain upper (Gastrointestinal disorders) | 8 | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 8 | 14
Weight decreased (Investigations) | 8 | 9
Insomnia (Psychiatric disorders) | 8 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 10
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 4
Dizziness (Nervous system disorders) | 7 | 2
Anaemia (Blood and lymphatic system disorders) | 7 | 3
Oedema peripheral (General disorders) | 5 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 8
Dry mouth (Gastrointestinal disorders) | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.